CLINICAL TRIAL: NCT04099771
Title: Low Dose Ketamine for Acute Management of Mood Disorders With Suicidal Ideation
Brief Title: Ketamine for Mood Disorders With Suicidal Ideation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1348833
Record Dates: First submitted 2019-06-14; First posted 2019-09-23 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorder, Major; Suicidal Ideation
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental): A total of 20 patients identified as having suicidal ideation will receive ketamine at 0.5mg/kg infused intravenously over 40 minutes.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine infusion

SUMMARY:
This study will explore whether the use of a medication, Ketamine, can help patients who come to the ER with thoughts of suicide by improving their mood and reducing thoughts of suicide. Ketamine has been used for this purpose in patients who have been hospitalized, but it has not been well studied in the ER. The investigators are first trying to show that patients and doctors in the ER find the treatment acceptable. The investigators also hope to determine whether Ketamine is effective in decreasing the severity of patient's suicidal thinking while in the ER. If this treatment works, future studies will look at whether it can help patients be discharged from the hospital earlier.

Research Procedures: Patients will be enrolled into the study on a voluntary basis after the research assistant has fully explained all the risks and benefits of the study (informed consent). Research assistants, Emergency Department staff, and the Psychiatry team will help identify patients for the study. Patients will be asked to complete surveys measuring the degree of their suicidal thinking and mood. Additional information will be collected on patients such as their demographics, current medications, and medical problems. Patients in the study will receive the medication, Ketamine, which will be given through an intravenous catheter (IV) at a dose based on the patient's weight and slowly infused over 40 minutes. Patients will be monitored during their stay in the Emergency Department by Emergency Department physicians and nurses for any signs of side effects to the medication. Patients will be asked to complete several surveys at specific time periods after the administration of Ketamine. All patients in the study will receive usual psychiatric care in addition to the study medication.

DETAILED DESCRIPTION:
Mood disorders complicated by suicidal ideation (SI) are common among patients presenting to the Emergency Department (ED). Under current standard practice, patients awaiting psychiatric evaluation in the emergency department do not typically receive interventions to address their mood disorder or SI. With no end to the extended ED boarding of psychiatric patients in sight, improvements in the acute treatment of SI with ketamine may help more patients receive prompt and appropriate treatment. Low-dose ketamine has been well studied in psychiatric literature. Studies involving a single dose of ketamine are promising, demonstrating both immediate and sustained reductions in suicidal ideations. Low dose ketamine has been well-studied in the ED for pain, asthma, and agitation, but not mood disorders or SI.

This study aims to determine whether or not it is feasible to administer low dose ketamine in the emergency department for the management of mood disorders with SI. Feasibility of ketamine administration in the ED and will be determined by: (1) ability to recruit participants, (2) tolerability of the intervention, and (3) acceptability by patients/providers. The investigators will also explore whether the administration of ketamine results in improvements in mood and SI.

This prospective open label feasibility pilot study will enroll 20 participants to receive ketamine at 0.5mg/kg infused intravenously over 40 minutes. Patients that have active suicidal ideation as determined by psychiatry staff who are being admitted to psychiatry under voluntary certification will be eligible for the study. The investigators will assess self-reported mood and suicidal ideations pre- and post-infusion of ketamine. Participants will complete assessments at baseline (pre-infusion), 2 hours and 6 hours post-infusion, and daily while in the ED until inpatient disposition.

The investigators hypothesize ketamine administration will be feasible in the emergency department and will result in improved mood and decreased SI.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* between 18 and 65 years of age
* have active suicidal ideation as determined by psychiatry staff
* are being admitted to psychiatry under voluntary certification and are able to provide informed consent.

Exclusion Criteria:

* have been previously enrolled in the trial
* are pregnant or breastfeeding; have a known or suspected allergy to ketamine; have used ketamine within 24h of presentation
* require antipsychotics (prescription or PRN by ED staff) or ED administration of other mood-altering medications for the management of acute agitation
* have known renal or liver failure; have neurologic, respiratory, or hemodynamic compromise as determined by the treating ED physician
* have history of stroke or cardiac disease (prior MI, cardiac stents or bypass surgery); or are incarcerated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and Rate of Participants Recruited into the Study throughout study period | One year
  The study will be considered feasible if the investigators are able to successfully enroll twenty participants into the study over a one year period (~1 - 2 participants per month).
Completion of total infusion of ketamine by participants | One year
  The study will be considered feasible if the intervention is tolerable to participants with no more than 25% of enrolled participants stopping the infusion of ketamine because of side effects (i.e., early stopping).
Percentage of participants and providers with positive response to ketamine administration | One year
  The study will be considered feasible if the intervention is considered acceptable to patients and providers (75% positive response on acceptability questionnaires).

SECONDARY OUTCOMES:
Reduction of SI in mood disorders by ketamine | 30 days
  The investigators will assess effectiveness based on changes in self-reported mood and suicidal ideations pre- and post-infusion of ketamine. Participants will complete assessments at baseline (pre-infusion), 2 hours and 6 hours post-infusion, and daily while in the ED until inpatient disposition. The investigators will use the assessments inherent rating scales to determine the reduction in SI, depression, or change in mood and determine if there was a significant decrease in SI in mood disorders after ketamine administration.

OTHER OUTCOMES:
Effect on in-patient length of stay | 30 days
  In exploratory analyses, the investigators will also examine a number of other outcomes including: the average length of stay of inpatient admission
Effect on indication of other medication administration | 30 days
  In exploratory analyses, the investigators will also examine concomitant medications received (e.g., for depression, agitation) by analyzing the percentage of patients who receive other medications in the emergency department.
Number of participants with return visit to the Emergency Department | 30 days
  In exploratory analyses, the investigators will also examine 30-day return ED visits via patient self-report and review of medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Beaudoin, MD PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States